CLINICAL TRIAL: NCT04583410
Title: Efficacy of Nicotine in Preventing COVID-19 Infection
Acronym: NICOVID-PREV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200538; 2020-003722-23 (EudraCT Number)
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Covid19; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere
Keywords: Covid19; SARS-COV2; Preventing infection
MeSH Terms: conditions — COVID-19 | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine patch (Experimental)
  Interventions: Drug: Nicotine patch
- Placebo patch (Placebo Comparator)
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Nicotine patch — NICOPATCHLIB, 7mg/24h Day 1 to day 3 : 3,5 mg/day Day 4 to day 9 : 7 mg/day Day 10 to Day 15 : 10,5 mg/day Day 16 to day 98 : 14 mg/day
  Decrease treatment Day 99 to day 105 : 10,5 mg/day Day 106 to day 112 : 7 mg/day Day 113 to Day 119 : 3,5 mg/day
  Arms: Nicotine patch
Drug: Placebo patch — PLACEBO OF NICOPATCHLIB, 7mg/24h Day 1 to day 3 : 3,5 mg/day Day 4 to day 9 : 7 mg/day Day 10 to Day 15 : 10,5 mg/day Day 16 to day 98 : 14 mg/day
  Decrease treatment Day 99 to day 105 : 10,5 mg/day Day 106 to day 112 : 7 mg/day Day 113 to Day 119 : 3,5 mg/day
  Arms: Placebo patch

SUMMARY:
The coronavirus disease (COVID-19) epidemic represents a major therapeutic challenge. The highly contagious severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) and the long duration of the disease have led to a massive influx of patients admitted in health services and intensive care units.

According to current knowledge, there are no treatments that prevent the spread of the infection, especially in exposed populations, or the disease progression to a severe form.

Daily active smokers are infrequent among outpatients or hospitalized patients with COVID-19. Several arguments suggest that nicotine is responsible for this protective effect via the nicotinic acetylcholine receptor (nAChR).

Nicotine may inhibit the penetration and spread of the virus and have a prophylactic effect in COVID-19 infection.

However, the epidemic is progressing throughout French territory and new variants (in particular the "English B1. 1.7 variant of SARS-COV-2") much more contagious run a risk of accelerating the epidemic in the population. The anti-SARS-COV-2 vaccines recently launched (or being evaluated) represent great hope in this health crisis, but trials were only able to show their effectiveness on symptomatic forms of SARS-COV-2 infection. On the one hand, the vaccination compaign for the entire population requires many months,which leaves many unprotected subjects waiting. In addition, there is currently no evidence of a protective role of vaccines against asymptomatic forms of COVID-19 and therefore on SARS-COV-2 transmission. Finally, the nicotine patches may protect people in hight-risk areas/periods until they are vaccinated (if they accept it and are eligible for it) and in the post-vaccination weeks necessary for the effectiveness of the vaccine,which reinforces the importance of evaluating this alternative prevention strategy, in the context of the arrival of vaccines

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. May be followed for the duration of the study
3. Obtaining free, informed and signed consent
4. Affiliated to a social security scheme or beneficiary of such a scheme (except AME)
5. Non-smoker and non-vaping (for former smokers or vapers: abstinent for at least 12 months)

Exclusion Criteria:

1. Symptoms suggestive of COVID-19 on the day of inclusion or in the past 14 days
2. Documented history of COVID-19 and / or positive SARS-COV2 serology before the day of inclusion
3. Treatment ongoing with nicotine replacement therapy, varenicline or bupropion within 30 days before inclusion
4. Known addiction problem to alcohol (defined by AUDIT-C > or = 10) or other substances.
5. Vaccinated against COVID19 infection.
6. Contraindications for nicotine patches:

   * pregnant woman (negative pregnancy test on inclusion) or breastfeeding woman
   * lack of effective contraception for women of childbearing potential
   * Generalized skin conditions that can interfere with the use of a transdermal patch
   * stroke or myocardial infarction or acute coronary syndrome for less than 3 months
   * allergy to nicotine or to one of the excipients of the transdermal patch
   * Uncontrolled high blood pressure
   * Unstable or worsening angor
   * Severe cardiac arrhythmia (defined by wearing an automatic implantable defibrillator)
   * Obliterating peripheral arterial disease
   * Known severe heart failure
   * Known severe renal or hepatic impairment,
   * Pheochromocytoma
   * Uncontrolled hyperthyroidism
   * Esophagitis due to gastroesophageal reflux disease or active peptic ulcer

     7 Already included in an interventional trial evaluating a health product 8 Staff under guardianship or curatorship or deprived of their liberty by a judicial or administrative decision 9 Do not have a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1633 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
SARS-COV2 seroconversion between W0 and W19 after randomization | Between week 0 and week 19
  This is the proportion of subjects with at least one positive serology between W2 and W19. The time of S19 takes into account a seroconversion delay of 5 weeks in relation to the SARS-CoV2 contamination.

SECONDARY OUTCOMES:
Proportion of documented symptomatic COVID-19 infection | Week 8, Week16
SARS-COV2 seroconversion | Week 16
  This is the proportion of patients with at least one positive serology between W2 and W16.
Asymptomatic COVID-19 infection proportion at week 14 | Week 14
  Asymptomatic COVID-19 infection is defined as SARS-CoV2 seroconversion at Week 19 without symptoms suggestive of COVID until the end of Week 16 to take in account of the two weeks of incubation period
Proportion of severe COVID-19 infection | Week 8, Week16
  documented infection (positive SARS-CoV2 PCR test and / or suggestive chest CT scan and / or seroconversion) whose first symptoms appeared before W8 and W16 respectively, and requiring hospitalization or home oxygen therapy, or having resulted in death
Number of sick leaves for a COVID-19 infection | Week 16
Number of days off during sick leaves for a COVID-19 infection | Week 16
Proportion of AE, SAE | From inclusion and week 25
Intensity and frequency of nausea, dizziness, feeling of empty head, headache, vomiting | Week 25
Proportion of active smoker or active vapers or taking nicotine substitutes documented by examination | Week 25
Proportion of active smoker or active vapers or taking nicotine substitutes documented by urinary cotinine | Week 25
Mean score of Desire to smoke defined by French Tobacco Craving scale | Week 25
Mean score of Withdrawal symptoms scale | Week 25
Dosage of cotinine in the urine | Week 8 and 25
Mean score of Fatigue Numeric rating scale | Week 2, week 8, week 16
Weight | Week 8, week 16, week 25
Mean score of Hospital anxiety and depression scale | Week 2, week 8, week 16
Mean score of Insomnia severity scale | Week 2, week 8, week 16
Positive and negative syndrome scale | Week 2, week 8, week 16

CONTACTS AND LOCATIONS:
Overall Officials: Zahir AMOURA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Centre Hospitalier Gonesse, Gonesse
  - Groupe Hospitalier de la Région de Mulhouse Sud Alsace, Mulhouse
  - Hôpital Pitié Salpêtrière - Service de Médecine Interne, Paris
  - Hôpital Sainte-Anne, Paris